CLINICAL TRIAL: NCT03211286
Title: Effect of Intravenous Tranexamic Acid on Reduction of Blood Losses in Hip Fracture Patients. A Randomized, Controlled, Double-blind Study
Brief Title: Effect of Intravenous Tranexamic Acid on Reduction of Blood Losses in Hip Fracture Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alejandro Lizaur-Utrilla, PhD, MD (Other)
Collaborators: University of Alicante (Other)
Responsible Party: Sponsor-Investigator, Alejandro Lizaur-Utrilla, PhD, MD, Head of Orthopaedic Surgery Department, Elda University Hospital
Organization: Elda University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TXA-Hip July2017
Record Dates: First submitted 2017-07-05; First posted 2017-07-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Hip Fractures; Anemia
Keywords: Hip fracture; Tranexamic acid; Perioperative blood loss; Blood Transfusion
MeSH Terms: conditions — Hip Fractures; Anemia | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: Patients will be treated surgically with a long trochanteric femoral nail (TFN) or hemiarthroplasty The two patient groups will include: 1) Study group treated with tranexamic acid at the time of surgical incision; 2) Control group treated with placebo injection (saline solution).
  Blood transfusion criteria will remain consistent with hospital standards. Deep vein thrombosis (DVT) prophylaxis will remain consistent with hospital standards (subcutaneous heparin from admission until 12 hours prior to surgery and beginning 6 hours after surgery). After discharge, .....
  Patients will be followed at regular intervals (1mo, 3mo, and at least 6mo) and at each time point the patient will be asked to report any adverse events (DVT, PT, Stroke, myocardial infarction, infection, hospitalization). Diagnostic studies to assess for thromboembolic events (i.e. DVT, pulmonary embolism (PE), and stroke) will be ordered only if the patient develops clinical signs or symptoms that justify their use.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be allocated into two groups based on randomized 20-block method by an independent assistant using computer generated randomization. Both patients and the treating surgeons will be blinded with regard to placebo vs. treatment until completion of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TXA group (Active Comparator): Tranexamic acid, a single dose of 1 g intravenous diluted in 100 mL saline solution at the time of surgical incision
  Interventions: Drug: Tranexamic Acid; Drug: Saline Solution
- Control group (Placebo Comparator): Saline solution, 100 mL intravenous at the time of surgical incision
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Tranexamic Acid — 1 g of intravenous tranexamic acid in 100 mL of saline solution
  Other Names: Saline solution
  Arms: TXA group
Drug: Saline Solution — saline solution 100 mL intravenous

SUMMARY:
Studies have shown that hip fractures have a significant perioperative blood loss. Postoperative anaemia is associated with a higher morbidity and mortality.

Tranexamic acid is a safe and effective antifibrinolytic widely used to reduce blood loss in other forms of orthopaedic surgery and in traumatized patients. However, evidence on the effectiveness of TXA in lower extremity fracture care is more limited.

Hip fractures represent a common orthopedic injury in a fragile patient population that often necessitates post-operative blood transfusion thereby putting the patient at additional risk of complications.

The goal of this study is to assess if the use of tranexamic acid in patients with hip fractures will result in a reduction in blood losses and blood transfusion rates.

Our hypothesis is that by providing intravenous TXA at the time of surgery will decrease the amount of preoperative and intraoperative bleeding thereby leading to a decreased need for postoperative transfusion.

This a double blinded, placebo controlled, therapeutic trial in which the patients will be randomized to receive TXA or a placebo (saline solution). Treatment will be administered pre-operatively as well as at the time of surgical incision. The primary outcome will be need for blood transfusion. Secondary outcomes will include calculated perioperative blood loss, length of stay, and rate of thromboembolic events, and 90 day mortality.

DETAILED DESCRIPTION:
Candidates for the study will be consecutive patients with a diagnosis of hip fractures treated at our center. All patients with hip fracture meeting inclusion criteria will be recruited for enrollment into the study. Informed consent will be obtained from the patient prior to randomization.

At that time, each patient will be randomized into one of two groups by a independent staff using computer generated randomization and allocation concealment. The two patient groups will include:

1. Study group: 1g of intravenous tranexamic acid at the time of surgical incision.
2. Control group: placebo injection (saline solution) at the time of surgical incision.

Both patients and the treating surgeons will be blinded with regard to placebo vs. treatment until completion of the study.

Patients will be treated surgically with a long trochanteric femoral nail (TFN) or hemiarthroplasty.

Blood transfusion criteria will remain consistent with hospital standards (Hb<8 g/dL or >9 g/dL if symptomatic anemia). Total number of blood transfusions received will be documented upon patient discharge.

Deep vein thrombosis (DVT) prophylaxis will remain consistent with hospital standards (subcutaneous heparin from admission until 12 hours prior to surgery and beginning 6 hours after surgery). After discharge, .....

Patients will be followed at regular intervals (1mo, 3mo, and at least 6mo) and at each time point the patient will be asked to report any adverse events (DVT, PT, Stroke, myocardial infarction, infection, hospitalization). Diagnostic studies to assess for thromboembolic events (i.e. DVT, pulmonary embolism (PE), and stroke) will be ordered only if the patient develops clinical signs or symptoms that justify their use.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients with a diagnosis of hip fractures treated at our hospital by any surgical procedureExclusion Criteria:
* Age over 60 years

Exclusion Criteria:

* ASA IV
* Concomitant fracture
* Refusal to receive blood products
* Preoperative anemia needing blood transfusion before surgery
* Severe comorbidity (cancer, severe pulmonary disease)
* Allergy for tranexamic acid.
* History of acute thromboembolic event (Deep Vein Thrombosis, Pulmonary Embolism, Stroke)
* Coagulopathy (INR > 1.4)
* Myocardial infarction in the previous 12 months
* Coronary stents
* Renal function impairment (serum creatinine > 2 mg/dL or creatinine clearance <30 mL/min),) or kidney transplant
* Platelet antiaggregant treatment in the week before surgery.
* Severe hepatic dysfunction (AST/ALT >60)
* History of hypercoagulability
* Acquired disturbances of color vision.
* Occurrence intraoperative surgical/medical/anesthetic complications

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
blood transfusion rate | Hospital stay, from admission to fourth day after surgery
  Number of patients needing blood transfusion

SECONDARY OUTCOMES:
Perioperative Blood Loss | Hospital stay, from admission to fourth day after surgery
  Measurement by serial hemoglobin and hematocrit, and calculation of loss by mathematical formulas
Infection rate | 90 postoperative days
  surgical and medical (pneumonia, urinary tract, etc)
Thrombotic events | 90 postoperative days
  Deep Venous Thrombosis, Pulmonary Embolism, Myocardial Infarction, Stroke
Mortality | 90 postoperative days
  number of deaths

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Lizaur-Utrilla, PHD, MD, Study Chair — Orthopaedic Surgery Department, Elda University Hospital
Locations (2):
- Spain (2):
  - Elda University Hospital, Elda, Alicante
  - Hospital Universitario de Elda, Elda, Alicante

IPD SHARING:
Plan to Share IPD: No